CLINICAL TRIAL: NCT06335823
Title: Randomized, Placebo-Controlled Study on the Efficacy of Transcutaneous Electrical Nerve Stimulation (TENS) for Pain Reduction During Intrauterine Device (IUD) Insertion in Outpatient Gynecology
Brief Title: Efficacy of Transcutaneous Electrical Nerve Stimulation (TENS) for Pain Reduction During Intrauterine Device (IUD) Insertion in Outpatient Gynecology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Jean Marino, APRN-CNP, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY20231621
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: IUD Insertion Pain
Keywords: contraception
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active TENS unit (Experimental): All patients will have the TENS unit applied: 2 pads from channel 1 will be at T10-L1 and the second set of pads will be from S2-S4; 5 minutes prior to the start of the procedure. Patients in this arm will have the TENS unit turned on to a 80 hz preset frequency with 100 mA as the pulse width.
  Interventions: Device: Transcutaneous electrical nerve stimulation (TENS)
- Non-active TENS unit (Placebo Comparator): All patients will have the TENS unit applied: 2 pads from channel 1 will be at T10-L1 and the second set of pads will be from S2-S4; 5 minutes prior to the start of the procedure. Patients will not have the TENS unit turned on.
  Interventions: Device: Placebo Transcutaneous electrical nerve stimulation (TENS)

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation (TENS) — All patients will have the TENS unit applied: 2 pads from channel 1 will be at T10-L1 and the second set of pads will be from S2-S4; 5 minutes prior to the start of the procedure. Patients will have the TENS unit turned on and half will have the TENS unit turned on to a 80 hz preset frequency with 100 mA as the pulse width.
  Arms: Active TENS unit
Device: Placebo Transcutaneous electrical nerve stimulation (TENS) — All patients will have the TENS unit applied: 2 pads from channel 1 will be at T10-L1 and the second set of pads will be from S2-S4; 5 minutes prior to the start of the procedure. Patients will have the TENS unit will not be turned on.
  Arms: Non-active TENS unit

SUMMARY:
Pain with intrauterine device (IUD) insertion is very common and there are few options for patients to help reduce this pain. Transcutaneous electric nerve stimulators (TENS) are a non-invasive procedure that may help reduce the pain with IUD insertions. The investigators hope that the information gleaned from this study will result in pain control options for future patients who desire an IUD placement.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years old
* Individuals with a cervix and uterus
* Seeking intrauterine device (IUD) placement for contraception or management of abnormal uterine bleeding
* Meet medical eligibility for IUD placement
* Ability to consent in English
* Ability to use the visual analogue scale (VAS)

Exclusion Criteria:

* Contraindications to IUD placement
* Use of analgesics within the last 4 hours prior to IUD placement
* Presence of a pacemaker

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Pain during IUD insertion as measured by the VAS score | IUD placement/introducer removal up to 5 minute
  The VAS score is a score of 0-10 with 0 being no pain and 10 being the worse pain imaginable

SECONDARY OUTCOMES:
Pain during IUD insertion as measured by the VAS score | speculum placement up to 1 minute
  The VAS score is a score of 0-10 with 0 being no pain and 10 being the worse pain imaginable
Pain during IUD insertion as measured by the VAS score | tenaculum placement up to 1 minute
  The VAS score is a score of 0-10 with 0 being no pain and 10 being the worse pain imaginable
Pain during IUD insertion as measured by the VAS score | sound insertion up to 5 minute
  The VAS score is a score of 0-10 with 0 being no pain and 10 being the worse pain imaginable
Pain during IUD insertion as measured by the VAS score | 5 minute post IUD insertion
  The VAS score is a score of 0-10 with 0 being no pain and 10 being the worse pain imaginable

OTHER OUTCOMES:
Pain during IUD insertion as measured by the VAS score | baseline
  The VAS score is a score of 0-10 with 0 being no pain and 10 being the worse pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Jean M Marino, APRN-CNP, Principal Investigator — University Hospitals
Locations (1):
- University Hospitals, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No